CLINICAL TRIAL: NCT06935409
Title: A Randomized, Controlled, Open-label, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of HS-20093 for Injection Versus Gemcitabine in Combination With Docetaxel in the Treatment of Osteosarcoma After Previous Second-line Treatment Failure (ARTEMIS-011)
Brief Title: Study of HS-20093 Versus Gemcitabine in Combination With Docetaxel in Treatment of Osteosarcoma After Previous Second-line Treatment Failure
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-304
Record Dates: First submitted 2025-04-17; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Osteosarcoma
Keywords: phase 3; osteosarcoma; HS-20093
MeSH Terms: conditions — Osteosarcoma | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HS-20093 (Experimental): Study participants in the experimental group shall continue to receive HS-20093 by intravenous infusion at a dose of 12.0 mg/kg, once every 3 weeks (Q3W) with a 21-day treatment cycle. Treatment shall continue until objective disease progression (excluding cases of treatment beyond PD or crossover treatment) or until other criteria for termination of study treatment specified in the protocol are met.
  Interventions: Drug: HS-20093
- Gemcitabine combined with docetaxel (Active Comparator): Study participants in the control arm will receive gemcitabine in combination with docetaxel. Gemcitabine (1000 mg/m2) will be administered intravenously over approximately 30 minutes on Days 1 and 8 of each 21-day treatment cycle, followed by docetaxel (75 mg/m2) on Day 8, intravenously over approximately 1 hour until objective disease progression or other criteria for treatment discontinuation are met.
  Interventions: Drug: Gemcitabine combined with docetaxel

INTERVENTIONS:
Drug: HS-20093 — Study participants in the experimental group shall continue to receive HS-20093 by intravenous infusion at a dose of 12.0 mg/kg, once every 3 weeks (Q3W) with a 21-day treatment cycle. Treatment shall continue until objective disease progression (excluding cases of treatment beyond PD or crossover treatment) or until other criteria for termination of study treatment specified in the protocol are met.
  Arms: HS-20093
Drug: Gemcitabine combined with docetaxel — Study participants in the control arm will receive gemcitabine in combination with docetaxel. Gemcitabine (1000 mg/m2) will be administered intravenously over approximately 30 minutes on Days 1 and 8 of each 21-day treatment cycle, followed by docetaxel (75 mg/m2) on Day 8, intravenously over approximately 1 hour until objective disease progression or other criteria for treatment discontinuation are met.
  Arms: Gemcitabine combined with docetaxel

SUMMARY:
This is a randomized, controlled, open, multicenter phase III clinical study to evaluate the efficacy and safety of HS-20093 for injection versus gemcitabine in combination with docetaxel in patients with osteosarcoma who have at least second-line treatment failure.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multicenter phase III clinical study to evaluate the efficacy and safety of HS-20093 for injection versus gemcitabine in combination with docetaxel in patients (≥ 12 years old) with osteosarcoma who have at least second-line treatment failure.

Eligible study participants shall be randomized in a 2:1 ratio to the experimental group and the control group. Study participants in the experimental group received HS-20093 at 12.0 mg/kg once every 3 weeks (Q3W), and the study participants continued to receive treatment until objective disease progression or other criteria for treatment discontinuation were met. Study participants in the control group received standard chemotherapy regimen of gemcitabine in combination with docetaxel until disease progression or other criteria for treatment discontinuation were met. The efficacy and safety of the two groups were evaluated after follow-up as per the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over 12 years old (≥ 12 years).
* Pathologically confirmed osteosarcoma (key IHC/tumor cell phenotyping results required for a definitive diagnosis must be provided).
* The study participants should have at least 1 target lesion based on RECIST 1.1.
* An ECOG PS of 0 to 1, with no exacerbation within two weeks prior to first dosing.
* A minimum expected survival of greater than 12 weeks.
* Female study participants of childbearing potential must be willing to use appropriate contraceptive measures and refrain from breastfeeding from the signing of informed consent to six months after the last dosing or the end of treatment (whichever occurs later); male study participants must be willing to use barrier contraceptive measures (i.e., condoms) from the signing of informed consent to six months after the last dosing or the end of treatment (whichever occurs later).
* Female study participants must provide negative blood or urine pregnancy test results within seven days before the first dosing, or meet one of the following criteria to prove there is no risk of pregnancy:
* Voluntary participation in this clinical trial, and signing and dating of the written ICF approved by the IRB/IEC in accordance with regulatory, local, and institutional guidelines.

Exclusion Criteria:

* Prior or ongoing therapies as follows:

  1. Prior or current use of treatments targeting B7-H3
  2. Prior or current use of treatments with topoisomerase I inhibitors, including antibody-drug conjugates that are effectively loaded with topoisomerase I inhibitors
  3. Prior or current use of systemic anti-tumor therapy with gemcitabine in combination with docetaxel;
  4. Use of cytotoxic chemotherapy drugs, experimental drugs, traditional Chinese medicines for anti-tumor indicationsor other anti-tumor drugs within 14 days prior to randomization; or requiring continued use of such drug therapies during the study;
  5. Use of macromolecular anti-tumor drug therapy within 28 days prior to randomization;
* Presence of residual grade ≥ 2 toxicities by Common Terminology Criteria for Adverse Events (CTCAE version 5.0) from previous treatments.
* History of other primary solid tumors.
* Inadequate bone marrow reserve or liver and kidney organ function, which meets any of the following laboratory limits:
* Serious, uncontrolled or active cardiovascular diseases.
* Severe or poorly controlled diabetes, including: ① Diabetic ketoacidosis or hyperglycemia and hyperosmolarity within 6 months prior to randomization; or ② other severe or poorly controlled diabetes conditions as determined by the investigator.
* Severe or poorly controlled hypertension, including: history of prior hypertensive crisis or hypertensive encephalopathy; adjustment of antihypertensive drug therapy within two weeks prior to randomization due to poor blood pressure control; systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg during the screening period.
* Have clinically significant hemorrhage symptoms or significant hemorrhagic diathesis within 1 month before randomization.
* Serious arteriovenous thrombotic events within 3 months before randomization, such as deep vein thrombosis, pulmonary embolism, etc. .
* Severe infection within four weeks prior to randomization, including but not limited to complications of infection, bacteremia, or severe pneumonia requiring intravenous antibiotic therapy for ≥ 2 weeks; or uncontrollable active infection during the screening period. Study participants who are receiving or have received prophylactic antibiotics may be enrolled.
* Patients who have received continuous glucocorticoid therapy for more than 30 days within 30 days before randomization, or who require long-term (≥ 30 days) use of glucocorticoids, or patients with other acquired/congenital immunodeficiency diseases or with a history of transplantation (except for corneal transplantation). Systemic corticosteroids (≤ 10 mg/d prednisone or equivalent) at a physiological replacement dose are permitted.
* Known presence of infectious diseases, such as hepatitis B , hepatitis C, tuberculosis , syphilis, or HIV infection , etc. Active infectious diseases will not be screened for proactively.
* Existing hepatic encephalopathy, hepatorenal syndrome, or ≥ Child-Pugh class B cirrhosis.
* Known interstitial pneumonia or immune pneumonitis, other moderate-to-severe lung diseases that may interfere with the detection or treatment of drug-related pulmonary toxicity and severely affect respiratory function.
* A history of prior serious neurological or psychiatric disorders, including epilepsy, dementia, severe depression, or other conditions that can interfere with the assessment.
* Female patients who are pregnant, breastfeeding, or planning to become pregnant during the study.
* Vaccination or occurrence of any degree of allergic or hypersensitivity reaction within four weeks prior to the first dosing.
* Subjects who have previously experienced severe allergies or serious infusion reactions, or who are allergic to recombinant humanized or murine protein substances.
* ‬Allergies to any component of the study drug HS-20093 , gemcitabine and its excipients, and docetaxel and its excipients.
* Patients who may have poor compliance with the study procedures and requirements as judged by the investigator.
* Patients with any condition that, in the Investigator's judgment, jeopardizes their safety or interferes with study assessments.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by IRC as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years.
  PFS is defined as the time interval from the randomization to disease progression as per ICR assessment or death due to any cause.

SECONDARY OUTCOMES:
ORR assessed by IRC as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years
  Confirmed ORR is defined as the sum of the complete response (CR) rate and partial response (PR) rate as per ICR per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
DCR assessed by IRC as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD (or non-CR/non-PD) per ICR per RECIST v1.1
DoR assessed by IRC as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) or death
ORR assessed by the investigator as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years
  Confirmed ORR is defined as the sum of the complete response (CR) rate and partial response (PR) rate as per investigator per RECIST v1.1
DCR assessed by the investigator as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD (or non-CR/non-PD) per investigator assessment per RECIST v1.1
DoR assessed by the investigator as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) or death
PFS assessed by the investigator as per RECIST 1.1 criteria | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 5 years
  PFS is defined as the time interval from the randomization to disease progression as per investigator assessment or death due to any cause
OS | From the date of randomization to the date of death due to any cause; Up to approximately 5 years
  Overall survival (OS) is defined as the time interval from randomization to death due to any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Jishuitan Hospital affiliated to Capital Medical University, Beijing
  - Peking University People's Hospital, Beijing